CLINICAL TRIAL: NCT01571297
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of RM-131 Administered to Patients With Diabetic Gastroparesis
Brief Title: Phase 2 Study to Evaluate Safety & Efficacy of RM-131 Administered to Patients With Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM-131-004
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus Complications; Gastroparesis
Keywords: Diabetes Mellitus; Delayed Gastric Emptying; Gastroparesis; Gastrointestinal Motility Disorder
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Gastroparesis | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RM-131 (Active Comparator)
  Interventions: Drug: RM-131
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-131 — Double blind RM-131 will be studied with various doses and regimens from 10 to 100 μg for 35 days.
  Arms: RM-131
Drug: Placebo — Placebo given subcutaneously for 35 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of RM-131 on gastric emptying, gastroparesis symptoms, and the safety and tolerability of RM-131 compared to placebo in patients with Type 1 and Type 2 diabetes mellitus and gastroparesis. The study is designed to evaluate the efficacy and safety of multiple dose regimens of RM-131. Study drug (RM-131 and placebo) will be administered subcutaneously in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to any study procedures and be willing and able to comply with study procedures.
* Type 1 or Type 2 diabetes mellitus with HbA1c ≤11% at screening.
* Diabetic gastroparesis defined as at least 3 months history of symptoms suggestive of gastroparesis on an ongoing basis.
* Average Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) > 2.6 during Visit 2.
* History of nausea and/or vomiting/emesis at least once a week during the 2 weeks prior to Visit 1.
* Delayed gastric emptying confirmed at screening by abnormal gastric emptying breath test (GEBT), defined as half-emptying time (t½) > 79 minutes.
* Stable concomitant medications defined as no changes in regimen for at least 2 weeks prior to Visit 2.
* No use of metoclopramide, erythromycin or anti-emetics for at least 2 weeks prior to Visit 2.
* Body mass index > 18 kg/m2.
* Female patients must have negative serum or urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. Female patients unable to bear children must have this documented in the electronic case report form (eCRF) (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]). Post-menopausal status will be confirmed by FSH.

Exclusion Criteria:

* Currently receiving parenteral feeding; presence of a nasogastric or other enteral tube for feeding or decompression.
* History of gastric surgery such as fundoplication, gastrectomy, gastric pacemaker placement, vagotomy, bariatric procedure.
* History of pyloric injection of botulinum toxin within 6 months of screening.
* Persistent daily vomiting.
* Patients with clinical suspicion of upper gastrointestinal obstruction must have been evaluated per standard of care, and obstruction ruled out before screening.
* Currently taking opiates.
* Currently taking GLP-1 and amylin analogs.
* Allergic or intolerant of egg, wheat, milk or algae, as these are components of the GEBT study meal.
* History of anorexia nervosa, binge-eating or bulimia within 5 years.
* ALT or AST > 2 X upper limit of normal during screening.
* History of intestinal malabsorption or pancreatic exocrine disease.
* Requires hemodialysis or has end-stage renal disease.
* History of human immunodeficiency virus (HIV) infection.
* Clinically significant neurologic or psychiatric disorders which are likely to impact compliance with protocol requirements.
* Poor venous access or inability to tolerate venipuncture.
* Participation in a clinical study within the 30 days prior to dosing in the present study.
* Any other reason, which in the opinion of the Investigator, including renal, hepatic or cardiopulmonary disease, or significant acute ECG abnormalities that would confound proper interpretation of the study or expose a patient to unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Effect of RM-131 on gastric emptying time | Screening and Day 28
  Change from baseline in gastric half-emptying time (t½)

SECONDARY OUTCOMES:
Effect of RM-131 on symptoms of gastroparesis | Baseline, daily for 28 days, and Day 35
  Longitudinal change from baseline over time in daily symptom scores from a self administered daily symptom diary
Safety and tolerability of RM-131 | From Screening through Day 35
  Assessment of adverse events and clinical laboratory evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Rhythm Pharmaceuticals, Inc.
Locations (30):
- United States (30):
  - Dothan, Alabama
  - Tucson, Arizona
  - North Little Rock, Arkansas
  - Concord, California
  - Lomita, California
  - Los Angeles, California
  - Torrance, California
  - Hialeah, Florida
  - Inverness, Florida
  - Miami, Florida
  - West Palm Beach, Florida
  - Wichita, Kansas
  - Monroe, Louisiana
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - Farmington Hills, Michigan
  - Jackson, Mississippi
  - Lebanon, New Hampshire
  - Albuquerque, New Mexico
  - Morehead City, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Dallas, Texas
  - Lubbock, Texas
  - Burke, Virginia
  - Norfolk, Virginia

REFERENCES:
- [Derived] Camilleri M, Lembo A, McCallum R, Tourkodimitris S, Kemps L, Miller MB, Bertelsen K, Iacob A. Overall safety of relamorelin in adults with diabetic gastroparesis: Analysis of phase 2a and 2b trial data. Aliment Pharmacol Ther. 2020 Jun;51(11):1139-1148. doi: 10.1111/apt.15711. Epub 2020 Apr 17. PMID 32301137
- [Derived] Lembo A, Camilleri M, McCallum R, Sastre R, Breton C, Spence S, White J, Currie M, Gottesdiener K, Stoner E; RM-131-004 Trial Group. Relamorelin Reduces Vomiting Frequency and Severity and Accelerates Gastric Emptying in Adults With Diabetic Gastroparesis. Gastroenterology. 2016 Jul;151(1):87-96.e6. doi: 10.1053/j.gastro.2016.03.038. Epub 2016 Apr 4. PMID 27055601